CLINICAL TRIAL: NCT06006312
Title: Establishment and Clinical Application of Pancreatic Endocrine and Exocrine Function Tests
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: SHDC12021107
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pancreatitis; Pancreatic Exocrine Insufficiency; Diabetes Mellitus; Community Populations; Fecal Elastase-1 Test
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Elderly population: The elderly population is defined as those over 60 years of age and residing in retirement home. Excluding people with critical conditions, mental disorders that prevent them from cooperating with the study, and those who are unable to defecate due to intestinal obstruction or other illnesses.
  Interventions: Diagnostic Test: fecal elastase-1 test
- Community population: This group is the resident population of the community. Excluding people with critical conditions, mental disorders that prevent them from cooperating with the study, and those who are unable to defecate due to intestinal obstruction or other illnesses.
  Interventions: Diagnostic Test: fecal elastase-1 test
- Chronic pancreatitis: Patients with chronic pancreatitis are considered as study subjects. If a CP patient has diabetes mellitus (exclude type 1 diabetes mellitus), a blood test will be performed to assess glycemic control.
  Interventions: Diagnostic Test: fecal elastase-1 test; Diagnostic Test: 72-hour fecal fat quantification; Diagnostic Test: blood sample test
- Type 2 diabetes mellitus: Patients with type 2 diabetes mellitus are considered as study subjects.
  Interventions: Diagnostic Test: fecal elastase-1 test; Diagnostic Test: blood sample test

INTERVENTIONS:
Diagnostic Test: fecal elastase-1 test — Personal information of the enrolled subjects will be collected and a fecal collection device will be distributed. Fecal elastase-1 levels will be measured after the fecal sample is collected.
Diagnostic Test: 72-hour fecal fat quantification — Enrolled subjects will eat a standard meal (100g of fat) daily for five consecutive days and collect stool samples for the last 72h. The fat content in the sample will be quantitatively detected and the fat absorption coefficient will be calculated.
  Groups: Chronic pancreatitis
Diagnostic Test: blood sample test — The enrolled subjects will undergo oral glucose tolerance test and will be collected blood samples for measurement of plasma glucose, insulin level, C-peptide level, glycosylated hemoglobin and vitamin.
  Other Names: oral glucose tolerance test
  Groups: Chronic pancreatitis; Type 2 diabetes mellitus

SUMMARY:
The goal of this observational study is to improve the epidemiological data of pancreatic exocrine insufficiency in China, determine the FE-1 cut-off value for the classification of PEI, and explore the characteristic differences between T3cDM and type 2 diabetes mellitus in clinical symptoms and laboratory indicators.

DETAILED DESCRIPTION:
Pancreatic exocrine insufficiency (PEI) refers to the reduction in the synthesis and secretion of pancreatic enzymes caused by various reasons, which leads to malabsorption and even nutritional deficiencies. The main causes of PEI include chronic pancreatitis (CP), acute pancreatitis, pancreatic cancer, pancreatectomy, enterectomy, diabetes mellitus and cystic fibrosis. Due to its numerous etiologies, the current prevalence of PEI is uncertain and very varied. The prevalence of PEI in the Chinese population is still lacking. Diagnosis of PEI in clinical practice is hindered by the lack of accurate tests, and it usually requires the combination of symptoms, nutritional markers and a noninvasive pancreatic function test in the appropriate clinical context. At present, the fecal elastase-1 (FE-1) test is the most widely applied non-invasive approach in routine clinical practice.

First, the study plans to record the baseline data of participants and perform the FE-1 test in specific elderly population and community population, in order to improve the epidemiology of PEI in China.

Second, the study will perform the FE-1 test in 100 CP patients, in order to determine the FE-1 cut-off value for the classification of PEI (mild-moderate and severe), using the coefficient of fat absorption as the "gold standard".

Third, people with CP often have diabetes mellitus which is described as type 3c diabetes mellitus (T3cDM). However, there are no recognized diagnostic criteria for T3cDM. Studies have shown that close to 50% of T3cDM cases are misclassified, most of which are diagnosed as type 2 diabetes mellitus (T2DM). According to certain research, the early stages of T3cDM are characterized by insufficient insulin and C-peptide secretion. The study will provide laboratory testing to 300 patients with T3cDM and T2DM in order to compare the differences and create T3cDM diagnostic criteria.

ELIGIBILITY:
For elderly population and community population:

Inclusion Criteria:

1. Agree to participate in the study and sign the informed consent.
2. Age of elderly participants are over 60 years old and the participants from community is unlimited.

Exclusion Criteria:

1. Participants in critical condition.
2. Have mental disorders and unable cooperate with investigators.
3. Have received bladder replacement with ileocolon surgery, or have intestinal obstruction and other diseases that can not defecate.

For chronic pancreatitis patients:

Inclusion Criteria:

1. Patients with chronic pancreatitis.
2. Age between 18 and 80 years.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Participants in critical condition.
3. Have mental disorders and unable cooperate with investigators.
4. Have received bladder replacement with ileocolon surgery, or have intestinal obstruction and other diseases that can not defecate.
5. Fecal sample quality, storage and transportation do not meet the requirements of fecal elastase-1 test.
6. Have undergone gastrectomy or pancreatectomy more than once.

For chronic pancreatitis patients with diabetes and patients with type 2 diabetes mellitus:

Inclusion Criteria (meet 1 or 2):

1. Patients with chronic pancreatitis and diabetes mellitus.
2. Patients with type 2 diabetes mellitus.

Exclusion Criteria:

1. Patients with type 2 diabetes mellitus.
2. Participants in critical condition.
3. Have mental disorders and unable cooperate with investigators.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Elderly participants will be recruited from several nursing homes. Community participants will be recruited from the community in Shanghai, China. Patients whti chronic pancreatitis and type 2 diabetes mellitus come from Changhai Hospital, Ruijin Hospital and Shanghai General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the prevalence of pancreatic exocrine insufficiency | 7 days after each participant collected stool samples
  Prevalence of pancreatic exocrine insufficiency (mild-moderate, sever) which is dependent on FE-1 level assessment in elderly population and community population respectively.

SECONDARY OUTCOMES:
Concentration of Glycosylated hemoglobin | 1 day after each participant collected blood sample
  Compare the concentration of glycosylated hemoglobin in chronic pancreatitis patients with diabetes mellitus and participants with type 2 diabetes mellitus.
Concentration of plasma glucose | 1 day after each participant collected blood sample
  During oral glucose tolerance test, concentration of plasma glucose (fasting and 2-hour) will be measured in chronic pancreatitis patients with diabetes mellitus and participants with type 2 diabetes mellitus.
C-peptide level | 1 day after each participant collected blood sample
  During oral glucose tolerance test, C-peptide levels (fasting and 2-hour) are measured in chronic pancreatitis patients with diabetes mellitus and participants with type 2 diabetes mellitus.
Insulin level | 1 day after each participant collected blood sample
  During oral glucose tolerance test, insulin levels (fasting and 2-hour) are measured in chronic pancreatitis patients with diabetes mellitus and participants with type 2 diabetes mellitus.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No